CLINICAL TRIAL: NCT05463835
Title: RubusElite Randomised Controlled Trial; Efficacy Testing of a Novel High Protein, Berry Polyphenol Enriched Dairy Beverage for Athletes and Physically Active Individuals
Brief Title: RubusElite Efficacy Testing of a Novel High Protein, Berry Polyphenol Enriched Dairy Beverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: South East Technological University (Unknown)
Responsible Party: Principal Investigator, Dr. Alice Lucey, Project Co-ordinator, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RubusEliteRCT
Record Dates: First submitted 2022-06-23; First posted 2022-07-19 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Muscle Damage; Muscle Soreness; Exercise Performance; Gut Microbiome; Stress; Anxiety
MeSH Terms: conditions — Myalgia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study will take the form of a 3-arm single blind parallel proof-of-concept RCT with two arms acting as active intervention arms and the third acting as a control arm. This study will use non-random convenience sampling. This sample will be obtained from a combination of sources including the WIT arena, the WIT student population as well being advertised on social media by the researcher, participants of local sporting clubs in the Southeast of Ireland who may be eligible may also be approached.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RubusElite dairy beverage (Experimental): The active treatment is a novel beverage, which has been formulated and developed by food Scientists at UCC. The RubusElite beverage is a science-led formulation of blackberry puree and high protein milk.
  Interventions: Dietary Supplement: RubusElite
- 'Protein rich' dairy beverage (Active Comparator): The high protein dairy beverage will be a commercially available high protein milk which is commercially produced.
  Interventions: Dietary Supplement: 'Protein rich' dairy beverage
- 'Low Protein' dairy beverage (Sham Comparator): The control beverage will be commercially available Taranis Dalia liquid commercially available low protein milk which will be purchased from the manufacturer for use in this study.
  Interventions: Dietary Supplement: 'Low Protein' dairy beverage

INTERVENTIONS:
Dietary Supplement: RubusElite — Each 500ml serving of this beverage will contain approximately 30g of milk protein alongside 750mg of polyphenols derived from blackberry puree. The study participant will consume 2 x 500ml per day which will contribute 60g protein and 1500mg polyphenols. No adverse effects associated with the consumption of dairy protein or berry fruits at the proposed intake levels have been reported to date.
  Arms: RubusElite dairy beverage
Dietary Supplement: 'Protein rich' dairy beverage — This dairy beverage will contain approximately 30g of milk protein /500ml serving and will not contain polyphenols.
  Arms: 'Protein rich' dairy beverage
Dietary Supplement: 'Low Protein' dairy beverage — This product also contains no polyphenols and negligible protein.
  Arms: 'Low Protein' dairy beverage

SUMMARY:
The RubusElite project is a multi-disciplinary project combining expertise in exercise science, nutrition, biochemistry, microbiology and food science across three institutions: University College Cork, Waterford Institute of Technology and Teagasc Food Research. This project has been funded by the Irish Department for Food, Agriculture and the Marines Food Institutional Research Measure (FIRM) initiative. The overarching aim of the RubusElite project is to provide an attractive, evidence-based performance and recovery food product for those undergoing frequent strenuous exercise in the form of a blackberry enriched, high protein dairy beverage. The process of developing this product will act as an exemplar model, providing best practice guidelines for the development of future functional foods in the performance nutrition space. This randomised controlled trial (RCT) will act as the ultimate test of efficacy of this functional food. It is envisaged that this RCT will assess the impact of a combined protein-polyphenol beverage on post-exercise recovery, exercise capacity, composition of the gut microbiome as well as central stress processing.

DETAILED DESCRIPTION:
This study will take the form of a 3-arm single blind parallel proof-of-concept RCT with two arms acting as active intervention arms and the third acting as a control arm. Prospective participants will be provided with a participant information sheet and informed consent form prior to any involvement in the protocol. It will be made clear to participants from the outset that their involvement in this study is entirely voluntary and they will be free to withdraw from the study at any point without having to provide any reason or explanation and without any risk of repercussions, either direct or indirect. Participants will receive a signed copy of their informed consent forms for their records. Once an initial interest has been expressed by a volunteer, they will be invited to complete an initial Eligibility Screening Form to assess their initial eligibility. If successful in meeting the initial criteria, participants will then be invited to the Human Performance Laboratory at WIT for an initial screening visit. Upon arrival to the laboratory participants will be provided with an opportunity to ask questions related to the information provided in the information sheet followed by signing the informed consent form. During the screening visit participants will be required to fill out a readiness to exercise form to ensure they are in adequate health to perform maximal exercise of the VO2peak test (Appendix 4). Once all inclusion and exclusion criteria are met and the participant is happy to proceed with their involvement in the study, they will then be scheduled to return to the laboratory to complete a baseline visit. During the baseline visit participants will provide a series of baseline fasted biological samples, alongside baseline psychological assessments and undertake a baseline 15km cycling time trial performance test.

Participants will be randomised to their assigned intervention arm at the end of their baseline visit and will be provided with a six-day supply of their randomised treatment beverage and will be instructed to consume two servings per day of this beverage (RubusElite beverage, high protein milk or low protein milk) for the following six days. On day 7, participants will return to the Human Performance Laboratory to complete a 'test exercise day' where they will undergo a repeat 15km cycling time trial performance test followed by a bout of unaccustomed drop-jump exercise consisting of 100 repetitions total. Participants will then be provided with a further 3-days of their treatment beverage and requested to return to the Human Performance Laboratory at 24h and 48h post-'test-exercise day' for follow-up assessment. Participants will also receive a 72h follow up phone call from the research team in order to assess muscular recovery post EIMD induction. Participants will be made aware that this call marks the end of their study participation, they will be thanked for their attendance and contribution to this research and will be notified of the overall study findings as soon as they are available.

This study will be conducted in accordance with Good Clinical Practice protocols, the research team will be appropriately qualified with sufficient training on such.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-45 Years of age • VO2peak between 35ml/kg/min and 55/ml/kg/min

Exclusion Criteria:

* Inability or unwillingness to discontinue use of any nutritional supplement or nutraceutical that may impact performance or recovery

  * Have an ongoing injury which will impact their ability to exercise, or a history of landing related lower limb injury
  * Being unwilling to consume a dairy product
  * Any diagnosis of a psychiatric disorder or taking any anti-psychotic, anxiolytic or anti-depressant medication
  * Any use of antibiotic medication within the previous two months or current use of prebiotic or probiotics.
  * Any diagnosis of chronic coexisting illness [cardiovascular, gastrointestinal (GI) [to include functional GI disorders, inflammatory bowel disease, coeliac disease, lactose intolerance]
  * Have a history of international sporting competition, or recent plyometric training

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Recovery of Maximal Isometric Mid-thigh Pull Strength | 48 hours post exercise
  Recovery of maximal muscle strength is assessed using an isometric mid-thigh pull following muscle damage inducing exercise. A fixed, immovable bar is set up at mid-thigh height directly above two force plates. While standing on the force plates the participant pulls on the bar as hard as possible for three continuous seconds and the maximal force produced is recorded in Newtons.
Recovery of Self-reported Muscle Soreness | 72 hours post exercise
  Self-reported muscle soreness is measured on a muscle pain scale ranging from 0 to 10. A score of 0 represents no pain at all while a sore of 10 represents extreme pain.
Recovery of Biomarkers of Oxidative Stress in Blood Plasma | 48 hours post exercise
  Oxidative stress measured by ELISA kit

SECONDARY OUTCOMES:
Time to Complete 15km Cycling Time Trial | 7 days
  The time taken to cycle 15km on a stationary bike is measured in minutes and seconds.
Heart Rate During 15km Cycling Time Trial | 7 days
  Heart rate is measured using a polar heart rate monitor at 5km, 10km and 15km during the 15km cycling time trial.
Average Power Output During 15km Cycling Time Trial | 7 days
  The average power output is measured in watts by the stationary bike throughout the 15km cycling time trial.
Blood Lactate Concentration in Blood During 15km Cycling Time Trial | 7 days
  Blood lactate is measured at 5km, 10km and 15km during the 15km cycling time trial. Blood is drawn from the earlobe and the blood lactate concentration is measured using a lactate pro meter.
Perceived Stress | 10 days
  Perceived stress is measured by Cohens self-report perceived stress scale. Scores range from 0 to 40. Scores from 0-13 represent low stress levels, 14-26 represent moderate stress and score greater than 26 represent high levels of stress.
Symptoms of Anxiety | 10 days
  Symptoms of anxiety are measured using the State Trait Anxiety Inventory. Scores for each of the forty items are summed giving a score ranging between 0 to 63. A score of 0 to 9 is normal, 10 to 18 is moderate anxiety, 19-29 is moderate to severe anxiety and a score above 29 is considered severe anxiety.
Depressive Symptoms | 10 days
  Depressive symptoms are measured using the Beck Depression Inventory II. Outcome scores range form 0 to 63. A score between 0 and 13 is considered minimal range, 14 to 19 is mild, 20 to 28 is moderate and above 28 is severe.
Gastrointestinal symptoms | 10 days
  Gastrointestinal symptoms are measured on line scales ranging from 0 to 100% where scores closer to 100% represent a negative outcome.
Positive and Negative Affect Schedule | 10 days
  Assessed using the Positive and Negative Affect Schedule self-report questionnaire. The scale comprises of twenty items. Ten of the items measure positive emotion and ten measure negative emotion. The ten items measuring positive emotion are summed giving a score ranging from 10 to 50 with 50 indicating more of a positive affect. The ten items measuring negative emotion are summed giving a score ranging from 10 to 50 with 50 indicating more of a negative affect.
Sleep Quality | 10 days
  Sleep quality is measured using the Pittsburgh Sleep Quality Index. The outcome is a score ranging from 0 to 21 with higher scores representing worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Doyle, PhD, Principal Investigator — Waterford Institute of Technology; Alice Lucey, PhD, Principal Investigator — University College Cork
Locations (1):
- Waterford Institute of Technology, Waterford, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No